CLINICAL TRIAL: NCT00291941
Title: A Multicentric, Randomised Study Comparing the Immunogenicity and Safety of Henogen's Adjuvanted Hepatitis B Vaccine Given at 0, 1, 6 Months to That of GSK Biologicals' Adjuvanted Hepatitis B Vaccine Given at 0, 1, 2, 6 Moths in Pre-Dialysis, and Dialysis Patients Who Are Hepatitis B Naive.
Brief Title: A Study to Compare the Immune Response and Safety Elicited by Henogen's Adjuvanted Hepatitis B Vaccine Compared to GSK Biologicals Adjuvanted Hepatitis B Vaccine in Pre-Dialysis and Dialysis Patients Who Have Not Been Exposed to Hepatitis B.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henogen (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sophie Houard CSO, Henogen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HN014/HBV-001 (105757); NCT00739726 (obsolete NCT alias)
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Hepatitis B
Keywords: Dialysis; Pre-dialysis; Hepatitis B vaccine; Prophylaxis
MeSH Terms: conditions — Hepatitis B | interventions — Fendrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Henogen HB vaccine
  Interventions: Biological: Henogen HBV vaccine
- 2 (Active Comparator): Fendrix vaccine
  Interventions: Biological: FENDRIX

INTERVENTIONS:
Biological: Henogen HBV vaccine — 20µg, Month 0, 2 and 6
  Arms: 1
Biological: FENDRIX — 20 µg,Months 0, 1, 2 and 6
  Arms: 2

SUMMARY:
The pre-dialysis, peritoneal dialysis and haemodialysis patients would benefit from an improved hepatitis B vaccine, which will elicit stronger and faster cellular and humoral immune responses after the primary vaccination course.

DETAILED DESCRIPTION:
Study participants will receive either Henogen's adjuvanted hepatitis B vaccine or GSK Biologicals' adjuvanted hepatitis B vaccine. The study involves a total of 7 visits and blood samples will taken at each of these visits.

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject 15 years of age or older at the time of the study entry.
* Written informed consent obtained from the subject/ from the parent or guardian of the subject.
* Seronegative for anti-HBs antibodies, anti-HBc antibodies and for HBsAg at screening.
* Pre-dialysis patients, peritoneal dialysis patients or haemodialysis patients.
* Non-childbearing potential female

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Use of any registered vaccine within 7 days before the first dose of study vaccine.
* Previous vaccination against hepatitis B (whether or not the subject responded to the vaccine).
* History of hepatitis B infection.
* Known exposure to hepatitis B virus within 6 months.
* Use of immunoglobulins within six months preceding the first study vaccination.
* Immunosuppression caused by the administration of parenteral steroids or chemotherapy (oral steroids are allowed).
* Any confirmed or suspected human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. oral/ axillary temperature < 37.5°C (or 37 °C in Czech Republic).
* Oral/axillary temperature superior or equal to 37.5°C (or 37 °C in Czech Republic).
* Pregnant or lactating female

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Anti-HBs seroprotection rate at Month 2. | Month 0 and 2

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | Months 0, 1, 2, 3, 6 and 7
Anti-HBs seroprotection rates for all subjects. | Months 0, 1, 2, 3, 6 and 7
Anti-HBs seropositivity rates for all subjects | Months 0, 1, 2, 3, 6 and 7
Percentage of subjects with anti-HBs antibody concentrations equal or greater than 100 mIU/ml for all subjects. | Months 0, 1, 2, 3, 6 and 7
Anti-HBs geometric mean concentrations calculated for all subjects. | Months 0, 1, 2, 3, 6 and 7
Anti-RF-1 seropositivity rates (defined as the percentage of subjects with anti-RF-1 like antibody concentrations superior or equal to 33 EU/ml, the assay cut-off) in a random subset of 50 subjects per group. | Months 0 and 7
Anti-RF-1 like antibody geometric mean concentration in a random subset of 50 subjects per group. | Month 0 and 7
Occurrence and intensity of solicited local signs and symptoms, as well as occurrence, intensity and relationship to vaccination of solicited general signs and symptoms during a 4-day follow-up (i.e. Day 0 to Day 3) after each vaccination and overall. | Month 0, 1, 2, 3, 6 and 7
Occurrence, intensity and relationship to vaccination of unsolicited symptoms reported during the 31-day (Day 0 to Day 30) follow-up period after each vaccination and overall. | Month 0, 1, 2, 3, 6 and 7
Occurrence, intensity and relationship to vaccination of all serious adverse events (SAEs) up to Month 7. | Month 0 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Christian Tielemans, MD, PhD, Principal Investigator — ULB Hôpital Erasme Département de Néphrologie
Locations (24):
- Belgium (14):
  - O.L.Vrouwziekenhuis Aalst, Aalst
  - RHMS La Madeleine ATH, Ath
  - RHMS Clinique Louis Caty Baudour, Baudour
  - AZ -VUB Dienst Nefrologie, Brussels
  - Cliniques universitaires Saint Luc, Brussels
  - CHU Brugmann (site V Horta) Service de néphrologie, Brussels
  - ULB Hôpital Erasme Département de Néphrologie, Brussels
  - CHU Hôpital civil de, Charleroi
  - UZ AntwerpenDienst nefrologie, Edegem
  - UZ Gent, Ghent
  - CHU Tivoli, La Louvière
  - UZ Gasthuisberg Leuven Nierziekten, Leuven
  - CHU Andre VESALE, Montigny-le-Tilleul
  - RHMS TournayService de néphrologie, Tournai
- Czechia (5):
  - Dept. of Heamodialysis Hospital JihlavaVrchlického, Jihlava
  - Regional Hospital Liberec, Liberec
  - Infection Diseases and AIDS Treatment ClinicUniversity Hospital with Outpatient Clinic, Ostrava - Poruba
  - Dept. of Internal Medicine StrahovSermirska 5, Prague
  - Masaryk´s Hospital Socialni pece 3316/12A, Ústí nad Labem
- Hungary (5):
  - St. Rókus Hospital, Budapest
  - St. István Hospital, Budapest
  - Petz Aladár Teaching Hospital Vasvári, Győr
  - Pest County Flór Ferenc Hospital, Kistarcsa
  - Vas and Szombathely County Markusovszky Hospital, Szombathely